CLINICAL TRIAL: NCT03177915
Title: Median Nerve Hydro-dissection Using Single Injection of Hyalase as a Novel Treatment of Carpal Tunnel Syndrome: Double Blind Randomized Clinical Trial
Brief Title: Median Nerve Hydro-dissection Using Single Injection of Hyalase as a Novel Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008406
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Carpal Tunnel Syndrome; Pain, Chronic
MeSH Terms: conditions — Carpal Tunnel Syndrome; Chronic Pain | interventions — hylase; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Investigate if, and to what extent, hydro-dissection using Hyalase versus saline, under ultrasound guidance, can improve the clinical condition, change in nerve conduction parameters of patients with CTS and delay or avoid the surgical intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyalase (Active Comparator): injection of Hyalase + 10 cc saline injection nearby median nerve as hydro-dissection
  Interventions: Drug: Hylase
- Saline (Active Comparator): Injection 10 cc saline injection as a median nerve hydro-dissection
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Hylase — median nerve hydro-dissection using Hyalase + 10 cc saline injection
  Other Names: ( group I )
  Arms: Hyalase
Drug: Saline — median nerve hydro-dissection using 10 cc saline injection
  Other Names: (group II)
  Arms: Saline

SUMMARY:
Carpal tunnel syndrome (CTS) is a common peripheral entrapment neuropathy, this study aims to investigate if, and to what extent hydro-dissection hyalase and saline of the median nerve could offer symptoms and clinical improvement

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common compression syndrome the upper extremities. Its problem has a high prevalence ranged estimated prevalence of 3.8% in the general population, 3 and 7.8% in the working population. It occurs at any age, especially in individuals in their 40s to 60s, and the male: female ratio is reported to be 3:7. A lot of treatment modalities have been tried to improve the condition, starting from local anesthetic injection, steroid, and up to surgical decompression of the nerves.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* complaining of carpal tunnel syndrome of 3 month duration or more
* diagnosed axonal neuropathy using electrodiagnosis , nerve conduction study

Exclusion Criteria:

* patient refusal infection at the site of intervention
* local anesthetic allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
pain alleviation | 6 months
  improvement of pain measured by visual analog scale , no pain the scale equal zero , and worst pain the scale equal 10

SECONDARY OUTCOMES:
Changes in ultrasound imaging | 6 months
  change of cross sectional area in cubic mellimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No